CLINICAL TRIAL: NCT04273256
Title: Myo-inositol for the Management of Poor Ovarian Responders: A Prospective Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Antoine Abou Moussa, professor of Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2018-0357
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Poor Ovarian Response
Keywords: Myo-inositol, In-vitro fertilization, Poor Ovarian Responders, Infertility
MeSH Terms: conditions — Infertility | interventions — Inositol

STUDY DESIGN:
Intervention Model Description: Upon consent, recruited women will be randomly allocated into either one of the study groups using a simple randomization method by computer-generated random numbers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myo-inositol arm (Experimental): Patients will be supplemented with 2 grams of Myo-inositol + at least 400 μg of folic acid (received from routinely prescribed multivitamins) every day for 3 months before the IVF cycle.
  Interventions: Drug: Myo-inositol
- Control arm (No Intervention): Patients will receive at least 400 μg of folic acid from routinely prescribed multivitamins every day for 3 months before the IVF cycle.

INTERVENTIONS:
Drug: Myo-inositol — patients who will be supplemented with 2 grams of Myo-inositol daily for 3 months prior to their in-vitro fertilization cycle
  Other Names: Celine
  Arms: Myo-inositol arm

SUMMARY:
The management of poor ovarian responders (POR) remains the most challenging in In-Vitro Fertilization (IVF). The incidence of POR ranges between 9 and 24% (Caprio F, et al, 2015).

POR refers to a reduction in the quantity of primordial follicle pool in reproductive age group (Jirge, P. R., 2016, Sunkara, S. K., et al, 2014), in addition to a higher risk of implantation failure (Kailasam C, et al, 2004).

To overcome this condition, fertility treatments using controlled ovarian stimulation along with IVF is needed to achieve pregnancy. Despite the use of various treatments including high dose gonadotropins, patients with POR have lower rates of pregnancy compared to patients with normal ovarian response (Oudendijk, J. F., et al, 2011). Studies now suggest a variety of regimens like the use of growth hormones, DHEA or androgens to improve the outcomes (Kyrou D, et al, 2009). The main interest of this study is the use of myo-inositol prior to IVF cycles for improvement of reproductive outcomes in poor ovarian responders.

DETAILED DESCRIPTION:
The management of poor ovarian responders (POR) remains the most challenging in In-Vitro Fertilization (IVF). The incidence of POR ranges between 9 and 24% (Caprio F, et al, 2015).

POR refers to a reduction in the quantity of primordial follicle pool in reproductive age group (Jirge, P. R., 2016, Sunkara, S. K., et al, 2014), in addition to a higher risk of implantation failure (Kailasam C, et al, 2004).

To overcome this condition, adjuvant fertility treatments using controlled ovarian stimulation along with IVF is needed to achieve pregnancy. Despite the use of various treatments including high dose gonadotropins, patients with POR have lower rates of pregnancy compared to patients with normal ovarian response (Oudendijk, J. F., et al, 2011). Studies now suggest a variety of regimens like the use of growth hormones, DHEA or androgens to improve the outcomes (Kyrou D, et al, 2009).

Inositol belongs to the vitamin B group, precursor for the synthesis of phosphatidylinositol polyphosphates (PIPs). PIPs belong to the signal transduction system involved in the regulation of different cellular functions such as signal transduction, cell morphogenesis and cytogenesis (Kutateladze TG, 2010). It is involved in cell membrane formation, lipid synthesis and cell growth (Unfer V, et al, 2012). It has been extensively studied in patients with insulin resistance, as inositol has an insulin sensitizing action (Croze ML & Soulage CO, 2013). In addition, researchers have hypothesized different mechanisms of action on different cell types especially at the level of the ovaries. An international consensus has confirmed that myo-inositol pre-treatment is able to improve the oocyte and the embryo quality via enhancing the intracellular Ca2+ oscillation with meiotic progression of germinal vesicle oocytes. Therefore, it acts on improving the oocyte maturation and embryo development (Nestler JE, et al, 1999, Papaleo E, et al, 2009).

Previous studies showed that higher concentrations of myo-inositol in follicular fluid are correlated with a better oocyte quality (Chiu TT, et al, 2002). A study by Jiang demonstrated that inositol supplementation reduces oxidative stress by different agents such as increasing superoxide dismutase and catalase levels (Jiang WD, et al, 2011). In view of its effects on oocyte maturation and quality, the use of myo-inositol in women with POR is promising. However, data is still sparse whether supplementation with myo-inostiol prior to IVF cycles does improve the pregnancy outcomes.

The main interest of this study is the use of myo-inositol prior to IVF cycles for improvement of reproductive outcomes in poor ovarian responders.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-44 years at the time of interview
* POR patients defined as: AMH<1.5 ng/nl, AFC of 7 or less, 5 oocytes or less retrieved in a previous cycle
* Patients undergoing controlled ovarian stimulation for any indication:

  * Male factor
  * Female factor

Exclusion Criteria:

* Patients with diabetes, thyroid dysfunction
* Patients with abnormal uterine cavity

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Retrieved oocytes | 4 months
  Number of oocytes retrieved (MII), including total number, number of mature MII, and proportion of dysmorphic oocytes

SECONDARY OUTCOMES:
Cycle cancellation rate | 4 months
  number of cycles cancelled before reaching embryo transfer
Fertilization rate | 4 months
  number of zygotes per number of oocytes inseminated
Implantation rate | 5 months
  number of intrauterine gestational sacs observed on transvaginal ultrasound divided by the number of transferred embryos
Clinical pregnancy rate per started treatment cycle (CPR) | 6 months
  the presence of a fetal heart beat on transvaginal ultrasound after 6-7 weeks of gestation
Ongoing pregnancy per embryo transferred | 7 months
  number of viable fetuses beyond 20 weeks' gestation per number of embryos transferred
Miscarriage rates | 7 months
  pregnancy loss prior to 12 weeks' gestation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Abu Mussa, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Background] Caprio F, D'Eufemia MD, Trotta C, Campitiello MR, Ianniello R, Mele D, Colacurci N. Myo-inositol therapy for poor-responders during IVF: a prospective controlled observational trial. J Ovarian Res. 2015 Jun 12;8:37. doi: 10.1186/s13048-015-0167-x. PMID 26067283
- [Background] Chiu TT, Rogers MS, Law EL, Briton-Jones CM, Cheung LP, Haines CJ. Follicular fluid and serum concentrations of myo-inositol in patients undergoing IVF: relationship with oocyte quality. Hum Reprod. 2002 Jun;17(6):1591-6. doi: 10.1093/humrep/17.6.1591. PMID 12042283
- [Background] Croze ML, Soulage CO. Potential role and therapeutic interests of myo-inositol in metabolic diseases. Biochimie. 2013 Oct;95(10):1811-27. doi: 10.1016/j.biochi.2013.05.011. Epub 2013 Jun 10. PMID 23764390
- [Background] Jirge PR. Poor ovarian reserve. J Hum Reprod Sci. 2016 Apr-Jun;9(2):63-9. doi: 10.4103/0974-1208.183514. PMID 27382229
- [Background] Jiang WD, Wu P, Kuang SY, Liu Y, Jiang J, Hu K, Li SH, Tang L, Feng L, Zhou XQ. Myo-inositol prevents copper-induced oxidative damage and changes in antioxidant capacity in various organs and the enterocytes of juvenile Jian carp (Cyprinus carpio var. Jian). Aquat Toxicol. 2011 Oct;105(3-4):543-51. doi: 10.1016/j.aquatox.2011.08.012. Epub 2011 Aug 27. PMID 21924699
- [Background] Kyrou D, Kolibianakis EM, Venetis CA, Papanikolaou EG, Bontis J, Tarlatzis BC. How to improve the probability of pregnancy in poor responders undergoing in vitro fertilization: a systematic review and meta-analysis. Fertil Steril. 2009 Mar;91(3):749-66. doi: 10.1016/j.fertnstert.2007.12.077. Epub 2008 Jul 21. PMID 18639875
- [Background] Kailasam C, Keay SD, Wilson P, Ford WC, Jenkins JM. Defining poor ovarian response during IVF cycles, in women aged <40 years, and its relationship with treatment outcome. Hum Reprod. 2004 Jul;19(7):1544-7. doi: 10.1093/humrep/deh273. Epub 2004 May 13. PMID 15142994
- [Background] Unfer V, Raffone E, Rizzo P, Buffo S. Effect of a supplementation with myo-inositol plus melatonin on oocyte quality in women who failed to conceive in previous in vitro fertilization cycles for poor oocyte quality: a prospective, longitudinal, cohort study. Gynecol Endocrinol. 2011 Nov;27(11):857-61. doi: 10.3109/09513590.2011.564687. Epub 2011 Apr 5. PMID 21463230
- [Background] Unfer V, Carlomagno G, Dante G, Facchinetti F. Effects of myo-inositol in women with PCOS: a systematic review of randomized controlled trials. Gynecol Endocrinol. 2012 Jul;28(7):509-15. doi: 10.3109/09513590.2011.650660. Epub 2012 Feb 1. PMID 22296306
- [Background] Papaleo E, Unfer V, Baillargeon JP, Fusi F, Occhi F, De Santis L. RETRACTED: Myo-inositol may improve oocyte quality in intracytoplasmic sperm injection cycles. A prospective, controlled, randomized trial. Fertil Steril. 2009 May;91(5):1750-1754. doi: 10.1016/j.fertnstert.2008.01.088. Epub 2008 May 7. PMID 18462730
- [Background] Oudendijk JF, Yarde F, Eijkemans MJ, Broekmans FJ, Broer SL. The poor responder in IVF: is the prognosis always poor?: a systematic review. Hum Reprod Update. 2012 Jan-Feb;18(1):1-11. doi: 10.1093/humupd/dmr037. Epub 2011 Oct 10. PMID 21987525
- [Background] Nestler JE, Jakubowicz DJ, Reamer P, Gunn RD, Allan G. Ovulatory and metabolic effects of D-chiro-inositol in the polycystic ovary syndrome. N Engl J Med. 1999 Apr 29;340(17):1314-20. doi: 10.1056/NEJM199904293401703. PMID 10219066